CLINICAL TRIAL: NCT01128738
Title: A Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled Study Including an Open-label Phase to Evaluate the Efficacy and Safety of GSK1358820 (Botulinum Toxin Type A) in Patients With Axillary Hyperhidrosis
Brief Title: GSK1358820 (Botulinum Toxin A) PhIII DB & OL Study in Patients With Axillary Hyperhidrosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 114078
Record Dates: First submitted 2010-05-20; First posted 2010-05-24 (Estimated); Results first posted 2012-04-25 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-05

CONDITIONS: Hyperhidrosis
Keywords: Neuromuscular Agents; Botulinum Toxin Type A; Sweating; Sweat Gland Disease; Axillary Hyperhidrosis; Skin Disease
MeSH Terms: conditions — Hyperhidrosis; Sweat Gland Diseases; Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK1358820 (Active Comparator): Onabotulinum toxin type A
  Interventions: Drug: GSK1358820
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK1358820 — Onabotulinum toxin type A
  Arms: GSK1358820
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The primary objective of this study is to demonstrate superiority of single treatment of GSK1358820 (hereinafter, referred to as BOTOX®) over placebo in terms of the efficacy of treatment with BOTOX® 50 U in each axilla (100 U in total for each patient) as intradermal injections based on gravimetric assessment (measurement of spontaneous axillary sweat production) for axillary hyperhidrosis.

ELIGIBILITY:
Inclusion Criteria:

<At start of the screening phase (Visit 1)>

* At least 50 mg of spontaneous resting axillary sweat production in each axilla measured gravimetrically at room temperature/humidity (20 - 25.6°C/20-80%) over a period of 5 minutes. (Patients should be at rest for at least 30 minutes after physical exercise including walking.)
* Patients with primary axillary hyperhidrosis whose excessive sweating in each axillae interferes daily life activities and whose Hyperhidrosis Disease Severity Scale (HDSS) score is 3 or 4.
* Age of 20 to 75 years at the time of informed consent.
* Both genders are eligible to enrol in the study. For men, only those who can practice contraception during the study period are eligible. Women of childbearing potential may be enrolled only if they have negative pregnancy test both in the screening period and just before treatment. Women of childbearing potential must agree to use one or more of the following reliable contraceptive measures throughout the study period:

  *: Abstinence, oral contraceptives, progesterone injection, levonorgestrel implant, estrogen ring, transdermal contraceptives, intrauterine device, vasectomized partner, and double-barrier contraception (condom or diaphragm with spermicidal jelly/film).
* QTc <450 msec, or QTc <480 msec in patients with bundle branch block. (QTc should be determined on one beat on echocardiogram (ECG) or determined by average on consecutive three beats.)
* Willing and able to provide written informed consent. <At start of the treatment phase (Visit 2)>
* At least 50 mg of spontaneous resting axillary sweat production in each axilla measured gravimetrically at room temperature/humidity (20 - 25.6°C/20-80%) over a period of 5 minutes. (Patients should be at rest for at least 30 minutes after physical exercise including walking.)
* Patients with primary axillary hyperhidrosis whose excessive sweating in each axillae interferes daily life activities and whose HDSS score is 3 or 4.
* Asparate aminotransferase (AST) and Alanine aminotransferase (ALT) < 2 x upper limit of normal (ULN), Alkaline phosphatase (ALP) and bilirubin <= 1.5 x ULN at Visit 1 (Free bilirubin >= 1.5 × ULN will not directly lead to study discontinuation if bilirubin fraction test result of direct bilirubin <35% is available.)

Exclusion Criteria:

<At start of the screening phase (Visit 1)>

* Any systemic neuromuscular junction disorder (e.g., myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis).
* Previous botulinum toxin treatment.
* Expected use of botulinum toxin for the treatment of any other disease during the study period.
* Known allergy to any of the components in the investigational product or iodine.
* Secondary hyperhidrosis, for example, hyperhidrosis that is secondary to other underlying diseases including hyperthyroidism, lymphoma and malaria.
* Previous surgical treatment of hyperhidrosis including sympathectomy, surgical debulking of the sweat glands, subcutaneous tissue curettage and ultrasonic surgery.
* Concurrent use of antibiotics that may interfere with neuromuscular junction function, for example, aminoglycoside antibiotics (e.g., gentamicin sulfate, fradiomycin sulfate), polypeptide antibiotics (e.g., polymixin B sulfate), tetracycline antibiotics, and lincomycin antibiotics, except for those contained in topical antimicrobials.
* Concurrent use of muscle relaxants (e.g., tubocurarin chloride hydrochloride hydrate, dantrolene sodium hydrate) or drugs that may have a muscle relaxant action (e.g. spectinomycin hydrochloride hydrate, antispasmogenics including baclofen, benzodiazepines and benzodiazepine-like drugs, benzamides).
* Chronic respiratory disorder.
* Serious muscle weakness or atrophy.
* Angle closure glaucoma or its precipitation (narrow angle).
* Dermal disorder including infection at anticipated injection sites in either axilla.
* Subject has serious physical symptom(s) (i.e., cardiac / hepatic / renal / hematopoietic disorder). The index of seriousness is Grade 3 of "criteria for classification of seriousness of adverse drug reactions to pharmaceutical products, etc. : Appendix 3" (Pharmaceutical Affairs bureau / Pharmaceutical and Chemical Safety Division (PAB / PSD) Notification No.80 in 1992).
* Anticipated need for surgery or hospitalization during the study period.
* Women who are pregnant, lactating, possibly pregnant or planning a pregnancy during the study period.
* Participation in another clinical study within 6 months of study entry or planned participation in another clinical study after entry to this study.
* Psychiatry disorder or cognitive disorder that may affect the patient's ability to give informed consent or to follow specified study procedures.
* History of alcohol or drug abuse.
* Any condition or situation that, in the investigator's or subinvestigator's opinion, may interfere with the patient's participation in the study.

<At start of the treatment phase (Visit 2)>

* Use of cholinomimetics, anticholinergics, antiperspirants containing aluminum chloride and deodorants, any oral herbal medicine treatments or any other topical treatments for hyperhidrosis within 7 days prior to study treatment..
* Underarm hair removed within 12 hours prior to study treatment or not removed sufficiently.
* Any condition or situation that, in the investigator's or subinvestigator's opinion, may interfere with the patient's participation in the study.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2010-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Japan (5):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Tokyo

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study consisted of a Screening Phase (1- to 2-week period), the First Treatment Phase (16- to 40-week period after first treatment), and the open-label Second Treatment Phase (16- to 24-week period after reinjection). All participants were observed until Week 40 after the first treatment irrespective of whether they received reinjection or not
Groups:
- BTX 50 U in First and Second TPs: Botulinum toxin type A (BTX) (GSK1358820) 50 units per axilla (underarm) (50 U/axilla) was injected intradermally to the hyperhidrotic area of both axillae at 10 to 15 injection sites during the First Treatment Phase (16- to 40-week period after first treatment). BTX 50 U/axilla was injected intradermally to the hyperhidrotic area of both axillae at 10 to 15 injection sites during the Second Treatment Phase (16- to 24-week period after reinjection). Participants who had a mean sweat production (measured by gravimetric assessment) in both axillae of beyond 50% of their Baseline (Week 0) level at any point in time during Weeks 16, 20, or 24 received a reinjection of BTX. Only participants who received this second treatment entered into the Second Treatment Phase.
- Placebo in First TP; BTX 50 U in Second TP: Placebo was injected intradermally to the hyperhidrotic area of both axillae at 10 to 15 injection sites during the First Treatment Phase. BTX 50 U/axilla was injected intradermally to the hyperhidrotic area of both axillae at 10 to 15 injection sites during the Second Treatment Phase. Participants who had a mean sweat production (measured by gravimetric assessment) in both axillae of beyond 50% of their Baseline (Week 0) level at any point in time during Weeks 16, 20, or 24 received an injection of BTX. Only participants who received this second treatment entered into the Second Treatment Phase.
Period: First Treatment Phase (TP)
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP
Started | 78 | 74
Completed | 74 | 73
Not Completed | 4 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 3 | 1
Period: Second TP
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP
Started | 34 (Only participants who received a second treatment entered this phase.) | 66 (Only participants who received a second treatment entered this phase.)
Completed | 34 | 63
Not Completed | 0 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP | Total
Number analyzed (Participants) | 78 | 74 | 152
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.2 (10.05) | 34.7 (11.69) | 35.5 (10.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 55 | 116
  Male | 17 | 19 | 36
Race/Ethnicity, Customized [Number; unit: participants]
  Asian-Japanese Heritage | 78 | 74 | 152

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders Assessed by Gravimetric Measurement at Week 4 in the First Treatment Phase
Description: A pre-weighed filter paper was placed into the axilla area to collect sweat over a 5-minute period. The paper was removed and weighed to determine the amount of sweat produced. A responder was defined as a participant showing at least a 50% reduction from Baseline in mean weight of axillary sweating.
Time Frame: Week 4
Population: Full Analysis Set for the First Treatment Phase (FAS1): all participants who received the first treatment of investigational product (IP) and had at least 1 post-Baseline efficacy assessment. The analysis was performed using the Last Observation Carried Forward (LOCF) dataset; missing data were imputed by carrying forward the last available data.
Measure: Number; unit: percentage of participants
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP
Number analyzed (Participants) | 78 | 74
percentage of participants | 96.2 | 45.9
Statistical Analysis 1: Comparison: BTX 50 U in First and Second TPs vs Placebo in First TP; BTX 50 U in Second TP; Test type: Superiority or Other; p < 0.001, Fisher Exact; Percentage difference = 50.2, 95% CI 2-sided [38.1 to 62.3] — Percentage difference was estimated as BTX 50 U minus placebo

2. Secondary Outcome: Percentage of Responders Assessed by Gravimetric Measurement at Weeks 1, 8, 12, 16, 20, and 24 in the First Treatment Phase
Description: as for outcome 1
Time Frame: Weeks 1, 8 ,12, 16, 20, and 24
Population: FAS1 (LOCF dataset). In the first treatment phase, the imputation of missing data by LOCF was performed up to Week 24; the missing data after Week 24 in the first treatment phase were not imputed.
Measure: Number; unit: percentage of participants
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP
Number analyzed (Participants) | 78 | 74
percentage of participants
  Week 1 | 93.6 | 52.7
  Week 8 | 94.9 | 48.6
  Week 12 | 89.7 | 62.2
  Week 16 | 87.2 | 32.4
  Week 20 | 74.4 | 20.3
  Week 24 | 56.4 | 9.5

3. Secondary Outcome: Mean Weight of Axillary Sweating by Gravimetric Measurement at Baseline and Weeks 1, 4, 8, 12, 16, 20, and 24 in the First Treatment Phase
Description: A pre-weighed filter paper was placed into the axilla area to collect sweat over a 5-minute period. The paper was removed and weighed to determine the amount of sweat produced.
Time Frame: Week 0 (Baseline); Weeks 1, 4, 8, 12, 16, 20, and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milligrams (mg)
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP
Number analyzed (Participants) | 78 | 74
milligrams (mg)
  Week 0 (Baseline) | 125.16 (85.366) | 137.45 (128.215)
  Week 1 | 17.58 (21.725) | 81.30 (117.296)
  Week 4 | 18.90 (36.500) | 82.92 (98.940)
  Week 8 | 15.47 (24.471) | 80.43 (121.172)
  Week 12 | 17.99 (28.380) | 68.31 (67.493)
  Week 16 | 18.60 (26.827) | 115.44 (157.710)
  Week 20 | 24.90 (31.793) | 127.30 (161.965)
  Week 24 | 44.27 (71.909) | 135.36 (159.123)

4. Secondary Outcome: Mean Percent Change From Baseline in Mean Weight of Axillary Sweating at Weeks 1, 4, 8, 12, 16, 20, and 24 in the First Treatment Phase
Description: A pre-weighed filter paper was placed into the axilla area to collect sweat over a 5-minute period. The paper was removed and weighed to determine the amount of sweat produced. Percent change from Baseline was calculated as follows: (mean weight at each visit minus mean weight at Baseline) * 100/mean weight at Baseline.
Time Frame: Week 0 (Baseline); and Weeks 1, 4, 8, 12, 16, 20, and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP
Number analyzed (Participants) | 78 | 74
percent change
  Week 1 | -82.4 (24.40) | -44.5 (53.32)
  Week 4 | -87.0 (16.00) | -34.3 (55.77)
  Week 8 | -84.8 (25.07) | -37.3 (51.64)
  Week 12 | -81.0 (37.10) | -33.6 (80.24)
  Week 16 | -78.8 (40.39) | -5.2 (109.55)
  Week 20 | -71.2 (43.99) | 1.9 (108.77)
  Week 24 | -55.6 (69.41) | 8.6 (105.13)

5. Secondary Outcome: Percentage of Responders Assessed by the Hyperhidrosis Severity Scale (HDSS) in the First Treatment Phase
Description: The HDSS is a 4-point scale (score range: 1-4) used to assess the impact of disease and the clinical relevance of treatment. Participants selected their underarm sweat condition from the following: 1=Never noticeable and never interferes with my daily activities, 2=Tolerable but sometimes interferes with my daily activities, 3=Barely tolerable and frequently interferes with my daily activities, and 4=Intolerable and always interferes with my daily activities. A responder was defined as a participant whose change from Baseline was equal to or less than -2.
Time Frame: Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, and 40
Population: FAS1. The number of participants remaining in the study at the time of the visit, particularly regardless of reinjection after Week 16, was used as the denominator. The number of participants analyzed varies by week because some participants were prematurely withdrawn or had no efficacy assessment at a particular time point.
Measure: Number; unit: percentage of participants
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP
Number analyzed (Participants) | 78 | 74
percentage of participants
  Week 1, n=78, 74 | 32.1 | 8.1
  Week 4, n=78, 73 | 61.5 | 13.7
  Week 8, n=78, 73 | 66.7 | 12.3
  Week 12, n=76, 73 | 57.9 | 13.7
  Week 16, n=76, 73 | 57.9 | 9.6
  Week 20, n=75, 73 | 48.0 | 9.6
  Week 24, n=76, 72 | 38.2 | 6.9
  Week 28, n=76, 71 | 36.8 | 4.2
  Week 32, n=74, 71 | 32.4 | 4.2
  Week 36, n=75, 70 | 30.7 | 4.3
  Week 40, n=74, 70 | 27.0 | 4.3

6. Secondary Outcome: Mean Change From Baseline in HDSS at Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, and 40 in the First Treatment Phase
Description: The HDSS is a 4-point scale (score range: 1-4) used to assess the impact of disease and the clinical relevance of treatment. Participants selected their underarm sweat condition from the following: 1=Never noticeable and never interferes with my daily activities, 2=Tolerable but sometimes interferes with my daily activities, 3=Barely tolerable and frequently interferes with my daily activities, and 4=Intolerable and always interferes with my daily activities. Change from Baseline in HDSS was calculated as follows: score at each visit minus score at Baseline.
Time Frame: Baseline and Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, and 40
Population: FAS1. The number of participants analyzed varies by week because some participants were prematurely withdrawn, had no efficacy assessment at a particular time point, or were entered into the Second Treatment Phase.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP
Number analyzed (Participants) | 78 | 74
scores on a scale
  Week 1, n=78, 74 | -1.1 (0.84) | -0.5 (0.71)
  Week 4, n=78, 73 | -1.6 (0.80) | -0.5 (0.84)
  Week 8, n=78, 73 | -1.7 (0.75) | -0.5 (0.77)
  Week 12, n=76, 73 | -1.6 (0.77) | -0.7 (0.80)
  Week 16, n=76, 73 | -1.6 (0.75) | -0.6 (0.71)
  Week 20, n=65, 24 | -1.6 (0.72) | -1.0 (0.78)
  Week 24, n=56, 15 | -1.6 (0.78) | -1.1 (0.88)
  Week 28, n=42, 6 | -1.7 (0.55) | -1.5 (0.55)
  Week 32, n=40, 7 | -1.6 (0.63) | -1.6 (0.79)
  Week 36, n=41, 7 | -1.6 (0.63) | -1.6 (0.79)
  Week 40, n=40, 7 | -1.5 (0.64) | -1.6 (0.79)

7. Secondary Outcome: Mean Change From Baseline in the Total Score of the Dermatology Life Quality Index (DLQI) at Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, and 40 in the First Treatment Phase
Description: The DLQI is a dermatology-specific, participant-answered questionnaire that allows for comparison of Quality of Life (QOL). DLQI total score (0-30) is a sum of the scores of 6 domains: Symptoms and Feelings, Daily Activities, Leisure, and Personal Relationships (score=0-6 for each); Work and School, and Treatment (score=0-3 for both; 0=not at all or not applicable, 3=very much or yes only in one item of Work and School). A lower score indicates better condition. Change from Baseline in the DLQI total score was calculated as follows: score at each visit minus score at Baseline.
Time Frame: Baseline and Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, and 40
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP
Number analyzed (Participants) | 78 | 74
scores on a scale
  Week 1, n=78, 74 | -5.4 (4.61) | -1.8 (3.49)
  Week 4, n=78, 73 | -6.6 (4.82) | -1.7 (3.66)
  Week 8, n=78, 73 | -6.9 (4.72) | -2.0 (3.89)
  Week 12, n=76, 73 | -6.9 (4.41) | -2.5 (4.26)
  Week 16, n=76, 73 | -6.9 (4.48) | -2.5 (4.25)
  Week 20, n=65, 24 | -6.7 (4.34) | -3.1 (4.37)
  Week 24, n=56, 15 | -6.9 (4.77) | -3.1 (4.53)
  Week 28, n=42, 6 | -7.3 (4.66) | -5.0 (4.73)
  Week 32, n=40, 7 | -7.1 (4.69) | -3.9 (6.47)
  Week 36, n=41, 7 | -6.9 (4.82) | -4.1 (5.70)
  Week 40, n=40, 7 | -6.5 (4.75) | -4.4 (5.19)

8. Secondary Outcome: Mean Change From Baseline in the Symptoms and Feelings Domain Score of the DLQI at Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, and 40 in the First Treatment Phase
Description: The DLQI is a dermatology-specific questionnaire that can be quickly answered by the participants and allows for comparison of QOL. The Symptoms and Feelings domain consists of 2 questions (Item 1 and Item 2). Scores range from 0 (not at all or not applicable) to 3 (very much) for each item; therefore, the possible total score for the Symptoms and Feelings domain is 0 to 6. A lower score indicates better condition. Change from Baseline in each domain score was calculated as follows: score at each visit minus score at Baseline.
Time Frame: Baseline and Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, and 40
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP
Number analyzed (Participants) | 78 | 74
scores on a scale
  Week 1, n=8, 74 | -0.9 (0.97) | -0.2 (0.95)
  Week 4, n=78, 73 | -1.2 (1.01) | -0.2 (0.90)
  Week 8, n=78, 73 | -1.3 (1.16) | -0.3 (0.87)
  Week 12, n=76, 73 | -1.3 (1.04) | -0.4 (0.96)
  Week 16, n=76, 73 | -1.3 (0.99) | -0.3 (1.04)
  Week 20, n=65, 24 | -1.2 (1.07) | -0.5 (1.06)
  Week 24, n=56, 15 | -1.3 (1.19) | -0.6 (1.06)
  Week 28, n=42, 6 | -1.5 (1.13) | -1.2 (0.98)
  Week 32, n=40, 7 | -1.4 (1.08) | -0.7 (1.50)
  Week 36, n=41, 7 | -1.3 (1.11) | -0.7 (1.50)
  Week 40, n=40, 7 | -1.3 (1.06) | -0.9 (1.21)

9. Secondary Outcome: Mean Change From Baseline in the Daily Activities Domain Score of the DLQI at Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, and 40 in the First Treatment Phase
Description: The DLQI is a dermatology-specific questionnaire that can be quickly answered by the participants and allows for comparison of QOL. The Daily Activities domain consists of 2 questions (Item 3 and Item 4). Scores range from 0 (not at all or not applicable) to 3 (very much) for each item; therefore, the possible total score for the Daily Activities domain is 0 to 6. A lower score indicates better condition. Change from Baseline in each domain score was calculated as follows: score at each visit minus score at Baseline.
Time Frame: Baseline and Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, and 40
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP
Number analyzed (Participants) | 78 | 74
scores on a scale
  Week 1, n=78, 74 | -1.8 (1.76) | -0.6 (1.40)
  Week 4, n=78, 73 | -2.2 (1.67) | -0.5 (1.33)
  Week 8, n=78, 73 | -2.4 (1.74) | -0.6 (1.44)
  Week 12, n=76, 73 | -2.4 (1.63) | -0.9 (1.45)
  Week 16, n=76, 73 | -2.4 (1.63) | -1.0 (1.38)
  Week 20, n=65, 24 | -2.3 (1.56) | -1.1 (1.35)
  Week 24, n=56, 15 | -2.4 (1.68) | -1.2 (1.57)
  Week 28, n=42, 6 | -2.5 (1.69) | -1.5 (1.52)
  Week 32, n=40, 7 | -2.4 (1.66) | -1.4 (1.62)
  Week 36, n=41, 7 | -2.4 (1.77) | -1.3 (1.38)
  Week 40, n=40, 7 | -2.1 (1.76) | -1.6 (1.62)

10. Secondary Outcome: Mean Change From Baseline in the Leisure Domain Score of the DLQI at Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, and 40 in the First Treatment Phase
Description: The DLQI is a dermatology-specific questionnaire that can be quickly answered by the participants and allows for comparison of QOL. The Leisure domain consists of 2 questions (Item 5 and Item 6). Scores range from 0 (not at all or not applicable) to 3 (very much) for each item; therefore, the possible total score for the Leisure domain is 0 to 6. A lower score indicates better condition. Change from Baseline in each domain score was calculated as follows: score at each visit minus score at Baseline.
Time Frame: Baseline and Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, and 40
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP
Number analyzed (Participants) | 78 | 74
scores on a scale
  Week 1, n=78, 74 | -1.4 (1.62) | -0.5 (1.37)
  Week 4, n=78, 73 | -1.6 (1.60) | -0.6 (1.33)
  Week 8, n=78, 73 | -1.7 (1.50) | -0.7 (1.38)
  Week 12, n=76, 73 | -1.7 (1.51) | -0.8 (1.45)
  Week 16, n=76, 73 | -1.7 (1.52) | -0.7 (1.45)
  Week 20, n=65, 24 | -1.7 (1.56) | -1.0 (1.53)
  Week 24, n=56, 15 | -1.9 (1.67) | -0.8 (1.52)
  Week 28, n=42, 6 | -1.8 (1.59) | -1.3 (1.63)
  Week 32, n=40, 7 | -1.8 (1.72) | -1.1 (2.19)
  Week 36, n=41, 7 | -1.7 (1.76) | -1.1 (2.19)
  Week 40, n=40, 7 | -1.7 (1.71) | -1.0 (1.91)

11. Secondary Outcome: Mean Change From Baseline in the Work and School Domain Score of the DLQI at Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, and 40 in the First Treatment Phase
Description: The DLQI is a dermatology-specific questionnaire that can be quickly answered by the participants and allows for comparison of QOL. The Work and School domain consists of 1 question (Item 7). The score for this item ranges from 0 (not at all or not applicable) to 3 (yes); therefore, the possible total score for the Work and School domain is 0 to 3. A lower score indicates better condition. Change from Baseline in each domain score was calculated as follows: score at each visit minus score at Baseline.
Time Frame: Baseline and Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, and 40
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP
Number analyzed (Participants) | 78 | 74
scores on a scale
  Week 1, n=78, 74 | -0.5 (0.64) | -0.2 (0.57)
  Week 4, n=78, 73 | -0.7 (0.75) | -0.1 (0.76)
  Week 8, n=78, 73 | -0.7 (0.79) | -0.1 (0.69)
  Week 12, n=76, 73 | -0.7 (0.79) | -0.2 (0.74)
  Week 16, n=76, 73 | -0.6 (0.78) | -0.1 (0.71)
  Week 20, n=65, 24 | -0.7 (0.73) | -0.3 (0.82)
  Week 24, n=56, 15 | -0.7 (0.78) | -0.2 (0.86)
  Week 28, n=42, 6 | -0.8 (0.73) | -0.5 (0.55)
  Week 32, n=40, 7 | -0.8 (0.66) | -0.1 (1.46)
  Week 36, n=41, 7 | -0.8 (0.82) | -0.4 (0.79)
  Week 40, n=40, 7 | -0.7 (0.65) | -0.6 (0.53)

12. Secondary Outcome: Mean Change From Baseline in the Personal Relationships Domain Score of the DLQI at Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, and 40 in the First Treatment Phase
Description: The DLQI is a dermatology-specific questionnaire that can be quickly answered by the participants and allows for comparison of QOL. The Personal Relationships domain consists of 2 questions (Item 8 and Item 9). Scores range from 0 (not at all or not applicable) to 3 (very much) for each item; therefore, the possible total score for the Personal Relationships domain is 0 to 6. A lower score indicates better condition. Change from Baseline in each domain score was calculated as follows: score at each visit minus score at Baseline.
Time Frame: Baseline and Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, and 40
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP
Number analyzed (Participants) | 78 | 74
scores on a scale
  Week 1, n=78, 74 | -0.4 (0.85) | -0.1 (0.61)
  Week 4, n=78, 73 | -0.4 (0.83) | -0.1 (0.64)
  Week 8, n=78, 73 | -0.4 (0.83) | -0.2 (0.68)
  Week 12, n=76, 13 | -0.4 (0.81) | -0.2 (0.80)
  Week 16, n=76, 73 | -0.4 (0.88) | -0.2 (0.84)
  Week 20, n=65, 24 | -0.4 (0.81) | -0.1 (0.74)
  Week 24, n=56, 15 | -0.4 (0.80) | -0.1 (0.70)
  Week 28, n=42, 6 | -0.4 (0.79) | -0.3 (0.82)
  Week 32, n=40, 7 | -0.4 (0.81) | -0.3 (0.76)
  Week 36, n=41, 7 | -0.4 (0.80) | -0.3 (0.76)
  Week 40, n=40, 7 | -0.4 (0.81) | -0.3 (0.76)

13. Secondary Outcome: Mean Change From Baseline in the Treatment Domain Score of the DLQI at Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, and 40 in the First Treatment Phase
Description: The DLQI is a dermatology-specific questionnaire that can be quickly answered by the participants and allows for comparison of QOL. The Treatment domain consists of 1 question (Item 10). The score for this item ranges from 0 (not at all or not applicable) to 3 (very much); therefore, the total possible score for the Treatment domain is 0 to 3. A lower score indicates better condition. Change from Baseline in each domain score was calculated as follows: score at each visit minus score at Baseline.
Time Frame: Baseline and Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, and 40
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP
Number analyzed (Participants) | 78 | 74
scores on a scale
  Week 1, n=78, 74 | -0.3 (0.65) | -0.1 (0.48)
  Week 4, n=78, 73 | -0.4 (0.69) | -0.1 (0.71)
  Week 8, n=78, 73 | -0.4 (0.69) | -0.2 (0.62)
  Week 12, n=76, 73 | -0.4 (0.62) | -0.1 (0.65)
  Week 16, n=76, 73 | -0.4 (0.66) | -0.1 (0.63)
  Week 20, n=65, 24 | -0.4 (0.63) | -0.1 (0.61)
  Week 24, n=56, 15 | -0.3 (0.69) | -0.2 (0.56)
  Week 28, n=42, 6 | -0.3 (0.64) | -0.2 (0.41)
  Week 32, n=40, 7 | -0.3 (0.56) | -0.1 (0.38)
  Week 36, n=41, 7 | -0.3 (0.57) | -0.3 (0.49)
  Week 40, n=40, 7 | -0.3 (0.64) | -0.1 (0.38)

14. Secondary Outcome: Mean Change From Baseline in the Item 1 (Itchy, Sore, Painful, or Stinging) Score of the DLQI at Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, and 40 in the First Treatment Phase
Description: The DLQI is a dermatology-specific questionnaire that can be quickly answered by the participants and allows for comparison of QOL. In Item 1, participants were asked how itchy, sore, painful or stinging their skin was over the last week. The scores for this item ranges from 0 (not at all or not applicable) to 3 (very much). Item 1 is in the Symptoms and Feelings domain. A lower score indicates better condition. Change from Baseline in each item score was calculated as follows: score at each visit minus score at Baseline.
Time Frame: Baseline and Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, and 40
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP
Number analyzed (Participants) | 78 | 74
scores on a scale
  Week 1, n=78, 74 | 0.0 (0.47) | 0.0 (0.39)
  Week 4, n=78, 73 | -0.1 (0.33) | 0.0 (0.33)
  Week 8, n=78, 73 | -0.1 (0.48) | 0.0 (0.46)
  Week 12, n=76, 73 | -0.1 (0.42) | -0.1 (0.40)
  Week 16, n=76, 73 | -0.1 (0.40) | 0.0 (0.39)
  Week 20, n=65, 24 | -0.1 (0.51) | 0.2 (0.38)
  Week 24, n=56, 15 | 0.0 (0.42) | 0.1 (0.26)
  Week 28, n=42, 6 | 0.0 (0.31) | 0.0 (0.00)
  Week 32, n=40, 7 | -0.1 (0.22) | 0.0 (0.00)
  Week 36, n=41, 7 | 0.0 (0.27) | 0.0 (0.00)
  Week 40, n=40, 7 | -0.1 (0.32) | 0.0 (0.00)

15. Secondary Outcome: Mean Change From Baseline in the Item 2 (Embarrassed or Self-Conscious) Score of the DLQI at Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, and 40 in the First Treatment Phase
Description: The DLQI is a dermatology-specific questionnaire that can be quickly answered by the participants and allows for comparison of QOL. In Item 2, participants were asked how embarrassed or self conscious they were because of their skin over the last week. The score for this item ranges from 0 (not at all or not applicable) to 3 (very much). Item 2 is in the Symptoms and Feelings domain. A lower score indicates better condition. Change from Baseline in each item score was calculated as follows: score at each visit minus score at Baseline.
Time Frame: Baseline and Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, and 40
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP
Number analyzed (Participants) | 78 | 74
scores on a scale
  Week 1, n=78, 74 | -0.9 (0.94) | -0.2 (0.92)
  Week 4, n=78, 73 | -1.1 (1.00) | -0.2 (0.87)
  Week 8, n=78, 73 | -1.2 (1.05) | -0.3 (0.85)
  Week 12, n=76, 73 | -1.2 (1.02) | -0.3 (0.91)
  Week 16, n=76, 73 | -1.2 (0.96) | -0.3 (0.94)
  Week 20, n=65, 24 | -1.2 (1.02) | -0.6 (0.92)
  Week 24, n=56, 15 | -1.3 (1.06) | -0.7 (0.98)
  Week 28, n=42, 6 | -1.4 (1.04) | -1.2 (0.98)
  Week 32, n=40, 7 | -1.4 (1.00) | -0.7 (1.50)
  Week 36, n=41, 7 | -1.3 (1.01) | -0.7 (1.50)
  Week 40, n=40, 7 | -1.2 (0.97) | -0.9 (1.21)

16. Secondary Outcome: Mean Change From Baseline in the Item 3 (Interfere Shopping/Caring for Home) Score of the DLQI at Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, and 40 in the First Treatment Phase
Description: The DLQI is a dermatology-specific questionnaire that can be quickly answered by the participants and allows for comparison of QOL. In Item 3, participants were asked how much their skin interfered with them going shopping or looking after their home or garden over the last week. The score for this item ranges from 0 (not at all or not applicable) to 3 (very much). Item 3 is in the Daily Activities domain. A lower score indicates better condition. Change from Baseline in each item score was calculated as follows: score at each visit minus score at Baseline.
Time Frame: Baseline and Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, and 40
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP
Number analyzed (Participants) | 78 | 74
scores on a scale
  Week 1, n=78, 74 | -0.6 (1.01) | -0.2 (0.77)
  Week 4, n=78, 73 | -0.8 (1.02) | -0.2 (0.76)
  Week 8, n=78, 73 | -0.8 (1.03) | -0.2 (0.75)
  Week 12, n=76, 73 | -0.8 (0.98) | -0.4 (0.89)
  Week 16, n=76, 73 | -0.8 (0.97) | -0.4 (0.86)
  Week 20, n=65, 24 | -0.8 (0.96) | -0.3 (0.75)
  Week 24, n=56, 15 | -0.8 (1.05) | -0.4 (0.91)
  Week 28, n=42, 6 | -0.9 (0.92) | -0.5 (0.84)
  Week 32, n=40, 7 | -0.9 (0.97) | -0.6 (0.79)
  Week 36, n=41, 7 | -0.9 (0.97) | -0.6 (0.79)
  Week 40, n=40, 7 | -0.8 (1.04) | -0.6 (0.79)

17. Secondary Outcome: Mean Change From Baseline in the Item 4 (Influenced Clothes You Wear) Score of the DLQI at Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, and 40 in the First Treatment Phase
Description: The DLQI is a dermatology-specific questionnaire that can be quickly answered by the participants and allows for comparison of QOL. In Item 4, participants were asked how much their skin interfered with the clothes they wore over the last week. The score for this item ranges from 0 (not at all or not applicable) to 3 (very much). Item 4 is in the Daily Activities domain. A lower score indicates better condition. Change from Baseline in each item score was calculated as follows: score at each visit minus score at Baseline.
Time Frame: Baseline and Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, and 40
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP
Number analyzed (Participants) | 78 | 74
scores on a scale
  Week 1, n=78, 74 | -1.2 (1.03) | -0.5 (0.88)
  Week 4, n=78, 73 | -1.5 (0.92) | -0.3 (0.90)
  Week 8, n=78, 73 | -1.6 (1.00) | -0.4 (1.01)
  Week 12, n=76, 73 | -1.6 (1.02) | -0.5 (0.90)
  Week 16, n=76, 73 | -1.6 (0.97) | -0.6 (0.91)
  Week 20, n=65, 24 | -1.5 (0.87) | -0.8 (0.78)
  Week 24, n=56, 15 | -1.5 (0.91) | -0.8 (1.08)
  Week 28, n=42, 6 | -1.6 (1.06) | -1.0 (0.89)
  Week 32, n=40, 7 | -1.5 (0.96) | -0.9 (1.21)
  Week 36, n=41, 7 | -1.5 (1.00) | -0.7 (1.11)
  Week 40, n=40, 7 | -1.3 (0.94) | -1.0 (1.15)

18. Secondary Outcome: Mean Change From Baseline in the Item 5 (Affected Social/Leisure Activities) Score of the DLQI at Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, and 40 in the First Treatment Phase
Description: The DLQI is a dermatology-specific questionnaire that can be quickly answered by the participants and allows for comparison of QOL. In Item 5, participants were asked how much their skin affected any social or leisure activities over the last week. The Score for this item ranges from 0 (not at all or not applicable) to 3 (very much). Item 5 is in the Leisure domain. A lower score indicates better condition. Change from Baseline in each item score was calculated as follows: score at each visit minus score at Baseline.
Time Frame: Baseline and Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, and 40
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP
Number analyzed (Participants) | 78 | 74
scores on a scale
  Week 1, n=78, 74 | -0.8 (0.94) | -0.2 (0.80)
  Week 4, n=78, 73 | -0.9 (0.92) | -0.3 (0.82)
  Week 8, n=78, 73 | -1.0 (0.92) | -0.3 (0.86)
  Week 12, n=76, 73 | -1.0 (0.94) | -0.4 (0.84)
  Week 16, n=76, 73 | -1.0 (0.95) | -0.4 (0.86)
  Week 20, n=65, 24 | -1.0 (0.93) | -0.3 (0.75)
  Week 24, n=56, 15 | -1.1 (0.97) | -0.1 (0.70)
  Week 28, n=42, 6 | -1.1 (0.98) | -0.5 (0.84)
  Week 32, n=40, 7 | -1.1 (1.02) | -0.4 (1.51)
  Week 36, n=41, 7 | -1.0 (1.02) | -0.4 (0.98)
  Week 40, n=40, 7 | -1.1 (0.99) | -0.4 (0.98)

19. Secondary Outcome: Mean Change From Baseline in the Item 6 (Difficult to Do Any Sport) Score of the DLQI at Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, and 40 in the First Treatment Phase
Description: The DLQI is a dermatology-specific questionnaire that can be quickly answered by the participants and allows for comparison of QOL. In Item 6, participants were asked how much their skin made it difficult to do any sports over the last week. The score for this item ranges from 0 (not at all or not applicable) to 3 (very much). Item 6 is in the Leisure domain. A lower score indicates better condition. Change from Baseline in each item score was calculated as follows: score at each visit minus score at Baseline.
Time Frame: Baseline and Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, and 40
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP
Number analyzed (Participants) | 78 | 74
scores on a scale
  Week 1, n=78, 74 | -0.6 (0.94) | -0.3 (0.85)
  Week 4, n=78, 73 | -0.7 (1.00) | -0.3 (0.85)
  Week 8, n=78, 73 | -0.7 (0.91) | -0.4 (0.86)
  Week 12, n=76, 73 | -0.7 (0.94) | -0.4 (0.91)
  Week 16, n=76, 73 | -0.7 (0.94) | -0.4 (0.90)
  Week 20, n=65, 24 | -0.7 (0.94) | -0.7 (1.16)
  Week 24, n=56, 15 | -0.7 (0.94) | -0.7 (1.10)
  Week 28, n=42, 6 | -0.7 (0.87) | -0.8 (0.98)
  Week 32, n=40, 7 | -0.7 (0.92) | -0.7 (0.95)
  Week 36, n=41, 7 | -0.7 (0.99) | -0.7 (1.38)
  Week 40, n=40, 7 | -0.7 (0.94) | -0.6 (1.13)

20. Secondary Outcome: Mean Change From Baseline in the Item 7 (Problem at Work or Studying) Score of the DLQI at Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, and 40 in the First Treatment Phase
Description: The DLQI is a dermatology-specific questionnaire that can be quickly answered by the participants and allows for comparison of QOL. In Item 7, participants were asked if their skin prevented them from working or studying over the last week. The score for this item ranges from 0 (not at all or not applicable) to 3 (yes). Item 7 is in the Work and School domain. A lower score indicates better condition. Change from Baseline in each item score was calculated as follows: score at each visit minus score at Baseline.
Time Frame: Baseline and Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, and 40
Population: FAS1 The number of participants analyzed varies by week because some participants were prematurely withdrawn, had no efficacy assessment at a particular time point, or were entered into the Second Treatment Phase.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP
Number analyzed (Participants) | 78 | 74
scores on a scale
  Week 1, n=78, 74 | -0.5 (0.64) | -0.2 (0.57)
  Week 4, n=78, 73 | -0.7 (0.75) | -0.1 (0.76)
  Week 8, n=78, 73 | -0.7 (0.79) | -0.1 (0.69)
  Week 12, n=76, 73 | -0.7 (0.79) | -0.2 (0.74)
  Week 16, n=76, 73 | -0.6 (0.78) | -0.1 (0.71)
  Week 20, n=65, 24 | -0.7 (0.73) | -0.3 (0.82)
  Week 24, n=56, 15 | -0.7 (0.78) | -0.2 (0.86)
  Week 28, n=42, 6 | -0.8 (0.73) | -0.5 (0.55)
  Week 32, n=40, 7 | -0.8 (0.66) | -0.1 (1.46)
  Week 36, n=41, 7 | -0.8 (0.82) | -0.4 (0.79)
  Week 40, n=40, 7 | -0.7 (0.65) | -0.6 (0.53)

21. Secondary Outcome: Mean Change From Baseline in the Item 8 (Problem With Partner/Friends) Score of the DLQI at Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, and 40 in the First Treatment Phase
Description: The DLQI is a dermatology-specific questionnaire that can be quickly answered by the participants and allows for comparison of QOL. In Item 8, participants were asked how much their skin created problems with their partner or any of their close friends or relatives over the last week. The score for this item ranges from 0 (not at all or not applicable) to 3 (very much). Item 8 is in the Personal Relationships domain. A lower score indicates better condition. Change from Baseline in each item score was calculated as follows: score at each visit minus score at Baseline.
Time Frame: Baseline and Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, and 40
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP
Number analyzed (Participants) | 78 | 74
scores on a scale
  Week 1, n=78, 74 | -0.3 (0.58) | -0.1 (0.42)
  Week 4, n=78, 73 | -0.3 (0.57) | -0.1 (0.45)
  Week 8, n=78, 73 | -0.3 (0.54) | -0.1 (0.51)
  Week 12, n=76, 73 | -0.3 (0.54) | -0.1 (0.55)
  Week 16, n=76, 73 | -0.3 (0.54) | -0.1 (0.60)
  Week 20, n=65, 24 | -0.3 (0.52) | -0.1 (0.41)
  Week 24, n=56, 15 | -0.3 (0.53) | -0.1 (0.46)
  Week 28, n=42, 6 | -0.3 (0.50) | -0.2 (0.41)
  Week 32, n=40, 7 | -0.3 (0.51) | -0.1 (0.38)
  Week 36, n=41, 7 | -0.2 (0.49) | -0.1 (0.38)
  Week 40, n=40, 7 | -0.3 (0.51) | -0.1 (0.38)

22. Secondary Outcome: Mean Change From Baseline in the Item 9 (Caused Any Sexual Difficulties) Score of the DLQI at Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36 and 40 in the First Treatment Phase
Description: The DLQI is a dermatology-specific questionnaire that can be quickly answered by the participants and allows for comparison of QOL. In Item 9, participants were asked how much their skin caused any sexual difficulties over the last week. The score for this item ranges from 0 (not at all or not applicable) to 3 (very much). Item 9 is in the Personal Relationships domain. A lower score indicates better condition. Change from Baseline in each item score was calculated as follows: score at each visit minus score at Baseline.
Time Frame: Baseline and Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, and 40
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP
Number analyzed (Participants) | 78 | 74
scores on a scale
  Week 1, n=78, 74 | -0.2 (0.40) | 0.0 (0.31)
  Week 4, n=78, 73 | -0.1 (0.39) | -0.1 (0.33)
  Week 8, n=78, 73 | -0.1 (0.42) | -0.1 (0.33)
  Week 12, n=76, 73 | -0.1 (0.39) | -0.1 (0.40)
  Week 16, n=76, 73 | -0.1 (0.47) | 0.0 (0.37)
  Week 20, n=65, 24 | -0.1 (0.39) | 0.0 (0.36)
  Week 24, n=56, 15 | -0.1 (0.41) | 0.0 (0.38)
  Week 28, n=42, 6 | -0.1 (0.40) | -0.2 (0.41)
  Week 32, n=40, 7 | -0.1 (0.40) | -0.1 (0.38)
  Week 36, n=41, 7 | -0.1 (0.40) | -0.1 (0.38)
  Week 40, n=40, 7 | -0.1 (0.40) | -0.1 (0.38)

23. Secondary Outcome: Mean Change From Baseline in the Item 10 (Problem Caused by Skin Treatment) Score of the DLQI at Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, and 40 in the First Treatment Phase
Description: The DLQI is a dermatology-specific questionnaire that can be quickly answered by the participants and allows for comparison of QOL. In Item 10, participants were asked how much of a problem the treatment for their skin was, for example, by making their home messy, or by taking up time. The Score for this item ranges from 0 (not at all or not applicable) to 3 (very much). Item 10 is in the Work and School domain. A lower score indicates better condition. Change from Baseline in each item score was calculated as follows: score at each visit minus score at Baseline.
Time Frame: Baseline and Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, and 40
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP
Number analyzed (Participants) | 78 | 74
scores on a scale
  Week 1, n=78, 74 | -0.3 (0.65) | -0.1 (0.48)
  Week 4, n=78, 73 | -0.4 (0.69) | -0.1 (0.71)
  Week 8, n=78, 73 | -0.4 (0.69) | -0.2 (0.62)
  Week 12, n=76, 73 | -0.4 (0.62) | -0.1 (0.65)
  Week 16, n=76, 73 | -0.4 (0.66) | -0.1 (0.63)
  Week 20, n=65, 24 | -0.4 (0.63) | -0.1 (0.61)
  Week 24, n=56, 15 | -0.3 (0.69) | -0.2 (0.56)
  Week 28, n=42, 6 | -0.3 (0.64) | -0.2 (0.41)
  Week 32, n=40, 7 | -0.3 (0.56) | -0.1 (0.38)
  Week 36, n=41, 7 | -0.3 (0.57) | -0.3 (0.49)
  Week 40, n=40, 7 | -0.3 (0.64) | -0.1 (0.38)

24. Secondary Outcome: Participant's Global Assessment of Treatment Satisfaction in the First Treatment Phase
Description: The participant's global assessment of treatment satisfaction is a method used to evaluate a participant's treatment satisfaction. Participants rated any improvement or worsening of their symptoms compared to Baseline by using the following 9-point scale: +4, Complete abolishment of signs and symptoms; +3, Marked improvement; +2, Moderate improvement; +1, Slight improvement; 0, Unchanged; -1, Slight worsening; -2, Moderate worsening; -3, Marked worsening; and -4, Very marked worsening.
Time Frame: Weeks 1, 4, 8, 12, 16, 20, 24, 28, 32, 36, and 40
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP
Number analyzed (Participants) | 78 | 74
scores on a scale
  Week 1, n=78, 74 | 1.8 (1.28) | 0.6 (0.95)
  Week 4, n=78, 73 | 2.6 (10.7) | 0.5 (1.05)
  Week 8, n=78, 73 | 2.7 (1.16) | 0.3 (0.96)
  Week 12, n=76, 73 | 2.6 (1.33) | 0.4 (0.86)
  Week 16, n=76, 73 | 2.6 (1.23) | 0.4 (0.83)
  Week 20, n=65, 24 | 2.6 (1.14) | 0.5 (1.06)
  Week 24, n=56, 15 | 2.5 (1.21) | 0.9 (1.22)
  Week 28, n=42, 6 | 2.9 (0.88) | 1.0 (1.26)
  Week 32, n=40, 7 | 2.6 (1.37) | 1.3 (1.38)
  Week 36, n=41, 7 | 2.5 (1.31) | 1.0 (1.63)
  Week 40, n=40, 7 | 2.4 (1.35) | 1.1 (1.46)

25. Secondary Outcome: Percentage of Responders Assessed by Gravimetric Measurement at Weeks 4, 8, 12, and 16 in the Second Treatment Phase
Description: A pre-weighed filter paper was placed into the axilla area to collect sweat over a 5-minute period. The paper was removed and weighed to determine the amount of sweat produced. A responder was defined as a participant showing at least a 50% reduction from Baseline (Week 0 in the Second Treatment Phase) in mean weight of axillary sweating.
Time Frame: Weeks 4 (Study Week 20 to 28), 8 (Study Week 24 to 32), 12 (Study Week 28 to 36), and 16 (Study Week 32 to 40) in the Second Treatment Phase
Population: FAS for the Second Treatment Phase (FAS2) (LOCF dataset): all participants who were included in the FAS1, received the second treatment of IP, and had at least one efficacy assessment after the second treatment. One participant who started the Second Treatment Phase was not included in the FAS2 because they had no efficacy assessment in this phase.
Measure: Number; unit: percentage of participants
Groups:
- Total: Total comprises all participants who received BTX 50 U/axillae in the Second Treatment Phase.
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP | Total
Number analyzed (Participants) | 34 | 65 | 99
percentage of participants
  Week 4 | 97.1 | 92.3 | 93.9
  Week 8 | 94.1 | 96.9 | 96.0
  Week 12 | 97.1 | 96.9 | 97.0
  Week 16 | 91.2 | 95.4 | 93.9

26. Secondary Outcome: Mean Weight of Axillary Sweating by Gravimetric Measurement at Baseline and Weeks 4, 8, 12, and 16 in the Second Treatment Phase
Description: as for outcome 3
Time Frame: Baseline (Week 0); Weeks 4 (Study Week 20 to 28), 8 (Study Week 24 to 32), 12 (Study Week 28 to 36), and 16 (Study Week 32 to 40) in the Second Treatment Phase
Population: FAS2 (LOCF dataset)
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP | Total
Number analyzed (Participants) | 34 | 65 | 99
mg
  Baseline (Week 0) | 84.50 (92.872) | 145.39 (163.635) | 124.48 (145.725)
  Week 4 | 6.69 (7.513) | 17.25 (35.386) | 13.62 (29.363)
  Week 8 | 11.37 (26.561) | 17.82 (36.049) | 15.61 (33.102)
  Week 12 | 15.22 (27.057) | 14.20 (20.411) | 14.55 (22.778)
  Week 16 | 12.87 (15.458) | 14.49 (21.217) | 13.94 (19.366)

27. Secondary Outcome: Mean Percent Change From Baseline in Mean Weight of Axillary Sweating at Weeks 4, 8, 12, and 16 in the Second Treatment Phase
Description: A pre-weighed filter paper was placed into the axilla area to collect sweat over a 5-minute period. The paper was removed and weighed to determine the amount of sweat produced. Percent change from Baseline in the Second Treatment phase was calculated as follows: (mean weight at each visit minus mean weight at Baseline in the Second Treatment Phase) * 100/mean weight at Baseline in the Second Treatment Phase.
Time Frame: Baseline (Week 0); and Weeks 4 (Study Week 20 to 28), 8 (Study Week 24 to 32), 12 (Study Week 28 to 36), and 16 (Study Week 32 to 40) in the Second Treatment Phase
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP | Total
Number analyzed (Participants) | 34 | 65 | 99
percent change
  Week 4 | -89.6 (15.20) | -84.6 (31.18) | -86.3 (26.80)
  Week 8 | -86.2 (16.76) | -84.4 (33.85) | -85.0 (29.04)
  Week 12 | -82.6 (18.43) | -87.6 (21.14) | -85.9 (20.30)
  Week 16 | -77.6 (32.23) | -84.5 (24.87) | -82.1 (27.65)

28. Secondary Outcome: Percentage of Responders Assessed by the HDSS in the Second Treatment Phase
Description: The HDSS is a 4-point scale (score range: 1-4) used to assess the impact of disease and the clinical relevance of treatment. Participants selected their underarm sweat condition from the following: 1=Never noticeable and never interferes with my daily activities, 2=Tolerable but sometimes interferes with my daily activities, 3=Barely tolerable and frequently interferes with my daily activities, and 4=Intolerable and always interferes with my daily activities. A responder was defined as a participant whose change from Baseline (Week 0 in the Second Treatment Phase) was equal to or less than -2.
Time Frame: Weeks 4 (Study Week 20 to 28), 8 (Study Week 24 to 32), 12 (Study Week 28 to 36), 16 (Study Week 32 to 40), 20 (Study Week 36 to 40), and 24 (Study Week 40) in the Second Treatment Phase
Population: FAS2. The number of participants analyzed varies by week because some participants were prematurely withdrawn or had no efficacy assessment at a particular time point.
Measure: Number; unit: percentage of participants
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP | Total
Number analyzed (Participants) | 34 | 65 | 99
percentage of participants
  Week 4, n=34, 65, 99 | 11.8 | 47.7 | 35.4
  Week 8, n=34, 65, 99 | 14.7 | 43.1 | 33.3
  Week 12, n=34, 64, 98 | 8.8 | 48.4 | 34.7
  Week 16, n=34, 62, 96 | 2.9 | 43.5 | 29.2
  Week 20, n=20, 56, 76 | 0 | 37.5 | 27.6
  Week 24, n=10, 49, 59 | 0 | 36.7 | 30.5

29. Secondary Outcome: Mean Change From Baseline in the HDSS at Weeks 4, 8, 12, 16, 20 and 24 in the Second Treatment Phase
Description: as for outcome 6
Time Frame: Baseline (Week 0) and Weeks 4 (Study Week 20 to 28), 8 (Study Week 24 to 32), 12 (Study Week 28 to 36), 16 (Study Week 32 to 40), 20 (Study Week 36 to 40), and 24 (Study Week 40) in the Second Treatment Phase
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP | Total
Number analyzed (Participants) | 34 | 65 | 99
scores on a scale
  Week 4, n=34, 65, 99 | -0.9 (0.61) | -1.5 (0.79) | -1.3 (0.79)
  Week 8, n=34, 65, 99 | -0.9 (0.65) | -1.4 (0.70) | -1.2 (0.72)
  Week 12, n=34, 64, 98 | -0.8 (0.64) | -1.4 (0.75) | -1.2 (0.77)
  Week 16, n=34, 62, 96 | -0.6 (0.54) | -1.3 (0.80) | -1.1 (0.78)
  Week 20, n=20, 56, 76 | -0.6 (0.51) | -1.2 (0.79) | -1.0 (0.77)
  Week 24, n=10, 49, 59 | -0.3 (0.67) | -1.1 (0.84) | -0.9 (0.86)

30. Secondary Outcome: Mean Change From Baseline in the Total Score of the DLQI at Weeks 4, 8, 12, 16, 20, and 24 in the Second Treatment Phase
Description: as for outcome 7
Time Frame: as for outcome 29
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP | Total
Number analyzed (Participants) | 34 | 65 | 99
scores on a scale
  Week 4, n=34, 65, 99 | -2.6 (2.65) | -4.0 (4.21) | -3.6 (3.79)
  Week 8, n=34, 65, 99 | -2.4 (3.18) | -4.0 (4.28) | -3.4 (4.00)
  Week 12, n=34, 64, 98 | -2.0 (2.72) | -3.9 (4.04) | -3.2 (3.74)
  Week 16, n=34, 62, 96 | -1.9 (2.48) | -3.7 (4.46) | -3.0 (3.96)
  Week 20, n=20, 56, 76 | -1.3 (1.41) | -3.3 (4.03) | -2.8 (3.63)
  Week 24, n=10, 49, 59 | -0.7 (3.20) | -3.3 (4.55) | -2.8 (4.43)

31. Secondary Outcome: Mean Change From Baseline in the Symptoms and Feelings Domain Score of the DLQI at Weeks 4, 8, 12, 16, 20, and 24 in the Second Treatment Phase
Description: as for outcome 8
Time Frame: as for outcome 29
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP | Total
Number analyzed (Participants) | 34 | 65 | 99
scores on a scale
  Week 4, n=34, 65, 99 | -0.5 (0.90) | -0.8 (0.86) | -0.7 (0.88)
  Week 8, n=34, 65, 99 | -0.6 (1.04) | -0.8 (0.89) | -0.8 (0.95)
  Week 12, n=34, 64, 98 | -0.5 (0.99) | -0.8 (0.84) | -0.7 (0.91)
  Week 16, n=34, 62, 96 | -0.4 (0.89) | -0.7 (0.93) | -0.6 (0.92)
  Week 20, n=20, 56, 76 | -0.3 (0.66) | -0.8 (0.84) | -0.6 (0.81)
  Week 24, n=10, 49, 59 | -0.1 (1.10) | -0.8 (0.85) | -0.7 (0.92)

32. Secondary Outcome: Mean Change From Baseline in the Daily Activities Domain Score of the DLQI at Weeks 4, 8, 12, 16, 20, and 24 in the Second Treatment Phase
Description: as for outcome 9
Time Frame: as for outcome 29
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP | Total
Number analyzed (Participants) | 34 | 65 | 99
scores on a scale
  Week 4, n=34, 65, 99 | -1.1 (1.07) | -1.4 (1.34) | -1.3 (1.26)
  Week 8, n=34, 65, 99 | -0.9 (1.08) | -1.3 (1.36) | -1.2 (1.28)
  Week 12, n=34, 64, 98 | -0.8 (1.06) | -1.3 (1.20) | -1.2 (1.17)
  Week 16, n=34, 62, 96 | -0.6 (1.07) | -1.2 (1.39) | -1.0 (1.31)
  Week 20, n=20, 56, 76 | -0.4 (0.82) | -1.0 (1.33) | -0.9 (1.25)
  Week 24, n=10, 49, 59 | -0.6 (1.07) | -1.1 (1.48) | -1.0 (1.42)

33. Secondary Outcome: Mean Change From Baseline in the Leisure Domain Score of the DLQI at Weeks 4, 8, 12, 16, 20, and 24 in the Second Treatment Phase
Description: as for outcome 10
Time Frame: as for outcome 29
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP | Total
Number analyzed (Participants) | 34 | 65 | 99
scores on a scale
  Week 4, n=34, 65, 99 | -0.6 (0.82) | -0.7 (0.97) | -0.6 (0.92)
  Week 8, n=34, 65, 99 | -0.4 (0.96) | -0.7 (1.02) | -0.6 (1.01)
  Week 12, n=34, 64, 98 | -0.4 (0.82) | -0.7 (1.03) | -0.6 (0.96)
  Week 16, n=34, 62, 96 | -0.5 (0.83) | -0.6 (1.01) | -0.6 (0.95)
  Week 20, n=20, 56, 76 | -0.3 (0.47) | -0.6 (0.89) | -0.5 (0.81)
  Week 24, n=10, 49, 59 | -0.2 (0.63) | -0.5 (1.02) | -0.5 (0.97)

34. Secondary Outcome: Mean Change From Baseline in the Work and School Domain Score of the DLQI at Weeks 4, 8, 12, 16, 20, and 24 in the Second Treatment Phase
Description: as for outcome 11
Time Frame: as for outcome 29
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP | Total
Number analyzed (Participants) | 34 | 65 | 99
scores on a scale
  Week 4, n=34, 65, 99 | -0.3 (0.51) | -0.6 (0.83) | -0.5 (0.75)
  Week 8, n=34, 65, 99 | -0.2 (0.65) | -0.5 (0.85) | -0.4 (0.80)
  Week 12, n=34, 64, 98 | -0.1 (0.56) | -0.5 (0.93) | -0.4 (0.83)
  Week 16, n=34, 62, 96 | -0.2 (0.43) | -0.5 (0.84) | -0.4 (0.74)
  Week 20, n=20, 56, 76 | -0.2 (0.37) | -0.4 (0.78) | -0.4 (0.71)
  Week 24, n=10, 49, 59 | -0.1 (0.57) | -0.4 (0.91) | -0.4 (0.87)

35. Secondary Outcome: Mean Change From Baseline in the Personal Relationships Domain Score of the DLQI at Weeks 4, 8, 12, 16, 20, and 24 in the Second Treatment Phase
Description: as for outcome 12
Time Frame: as for outcome 29
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP | Total
Number analyzed (Participants) | 34 | 65 | 99
scores on a scale
  Week 4, n=34, 65, 99 | -0.1 (0.29) | -0.3 (0.77) | -0.2 (0.65)
  Week 8, n=34, 65, 99 | 0.0 (0.30) | -0.3 (0.81) | -0.2 (0.69)
  Week 12, n=34, 64, 98 | -0.1 (0.29) | -0.3 (0.78) | -0.2 (0.66)
  Week 16, n=34, 62, 96 | 0.0 (0.30) | -0.3 (0.89) | -0.2 (0.75)
  Week 20, n=20, 56, 76 | 0.0 (0.30) | -0.3 (0.73) | -0.2 (0.63)
  Week 24, n=10, 49, 59 | 0.2 (0.63) | -0.3 (0.87) | -0.2 (0.85)

36. Secondary Outcome: Mean Change From Baseline in the Treatment Domain Score of the DLQI at Weeks 4, 8, 12, 16, 20, and 24 in the Second Treatment Phase
Description: as for outcome 13
Time Frame: as for outcome 29
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP | Total
Number analyzed (Participants) | 34 | 65 | 99
scores on a scale
  Week 4, n=34, 65, 99 | -0.1 (0.50) | -0.3 (0.59) | -0.2 (0.56)
  Week 8, n=34, 65, 99 | -0.1 (0.36) | -0.3 (0.62) | -0.2 (0.55)
  Week 12, n=34, 64, 98 | 0.0 (0.30) | -0.3 (0.60) | -0.2 (0.52)
  Week 16, n=34, 62, 96 | -0.1 (0.29) | -0.2 (0.73) | -0.2 (0.62)
  Week 20, n=20, 56, 76 | -0.1 (0.31) | -0.2 (0.69) | -0.2 (0.61)
  Week 24, n=10, 49, 59 | 0.1 (0.32) | -0.2 (0.73) | -0.1 (0.68)

37. Secondary Outcome: Mean Change From Baseline in the Item 1 (Itchy, Sore, Painful, or Stinging) Score of the DLQI at Weeks 4, 8, 12, 16, 20, and 24 in the Second Treatment Phase
Description: The DLQI is a dermatology-specific questionnaire that can be quickly answered by the participants and allows for comparison of QOL. In Item 1, participants were asked how itchy, sore, painful or stinging their skin was over the last week. The score for this item ranges from 0 (not at all or not applicable) to 3 (very much). Item 1 is in the Symptoms and Feelings domain. A lower score indicates better condition. Change from Baseline in each item score was calculated as follows: score at each visit minus score at Baseline.
Time Frame: as for outcome 29
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP | Total
Number analyzed (Participants) | 34 | 65 | 99
scores on a scale
  Week 4, n=34, 65, 99 | -0.1 (0.55) | -0.1 (0.30) | -0.1 (0.40)
  Week 8, n=34, 65, 99 | -0.1 (0.56) | -0.1 (0.35) | -0.1 (0.43)
  Week 12, n=34, 64, 98 | -0.1 (0.56) | 0.0 (0.38) | -0.1 (0.45)
  Week 16, n=34, 62, 96 | -0.1 (0.50) | 0.0 (0.40) | -0.1 (0.44)
  Week 20, n=20, 56, 76 | -0.1 (0.51) | -0.1 (0.32) | -0.1 (0.38)
  Week 24, n=10, 49, 59 | 0.1 (0.57) | -0.1 (0.31) | -0.1 (0.37)

38. Secondary Outcome: Mean Change From Baseline in the Item 2 (Embarrassed or Self-conscious) Score of the DLQI at Weeks 4, 8, 12, 16, 20, and 24 in the Second Treatment Phase
Description: as for outcome 15
Time Frame: as for outcome 29
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP | Total
Number analyzed (Participants) | 34 | 65 | 99
scores on a scale
  Week 4, n=34, 65, 99 | -0.4 (0.66) | -0.8 (0.79) | -0.6 (0.76)
  Week 8, n=34, 65, 99 | -0.5 (0.71) | -0.8 (0.81) | -0.7 (0.78)
  Week 12, n=34, 64, 98 | -0.3 (0.84) | -0.7 (0.76) | -0.6 (0.81)
  Week 16, n=34, 62, 96 | -0.3 (0.67) | -0.7 (0.83) | -0.5 (0.79)
  Week 20, n=20, 56, 76 | -0.3 (0.44) | -0.7 (0.81) | -0.6 (0.75)
  Week 24, n=10, 49, 59 | -0.2 (0.63) | -0.7 (0.85) | -0.6 (0.83)

39. Secondary Outcome: Mean Change From Baseline in the Item 3 (Interfere Shopping/Caring for Home) Score of the DLQI at Weeks 4, 8, 12, 16, 20, and 24 in the Second Treatment Phase
Description: as for outcome 16
Time Frame: as for outcome 29
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP | Total
Number analyzed (Participants) | 34 | 65 | 99
scores on a scale
  Week 4, n=34, 65, 99 | -0.3 (0.47) | -0.4 (0.60) | -0.4 (0.56)
  Week 8, n=34, 65, 99 | -0.3 (0.57) | -0.3 (0.59) | -0.3 (0.58)
  Week 12, n=34, 64, 98 | -0.3 (0.51) | -0.3 (0.49) | -0.3 (0.50)
  Week 16, n=34, 62, 96 | -0.3 (0.51) | -0.3 (0.57) | -0.3 (0.55)
  Week 20, n=20, 56, 76 | -0.2 (0.41) | -0.3 (0.65) | -0.3 (0.60)
  Week 24, n=10, 49, 59 | -0.4 (0.52) | -0.3 (0.60) | -0.3 (0.59)

40. Secondary Outcome: Mean Change From Baseline in the Item 4 (Influenced Clothes You Wear) Score of the DLQI at Weeks 4, 8, 12, 16, 20, and 24 in the Second Treatment Phase
Description: as for outcome 17
Time Frame: as for outcome 29
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP | Total
Number analyzed (Participants) | 34 | 65 | 99
scores on a scale
  Week 4, n=34, 65, 99 | -0.7 (0.71) | -1.0 (0.93) | -0.9 (0.87)
  Week 8, n=34, 65, 99 | -0.6 (0.69) | -1.0 (0.93) | -0.8 (0.86)
  Week 12, n=34, 64, 98 | -0.6 (0.66) | -1.0 (0.89) | -0.9 (0.85)
  Week 16, n=34, 62, 96 | -0.4 (0.70) | -0.9 (1.03) | -0.7 (0.96)
  Week 20, n=20, 56, 76 | -0.2 (0.52) | -0.8 (0.94) | -0.6 (0.88)
  Week 24, n=10, 49, 59 | -0.2 (0.63) | -0.8 (1.08) | -0.7 (1.04)

41. Secondary Outcome: Mean Change From Baseline in the Item 5 (Affected Social/Leisure Activities) Score of the DLQI at Weeks 4, 8, 12, 16, 20, and 24 in the Second Treatment Phase
Description: as for outcome 18
Time Frame: as for outcome 29
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP | Total
Number analyzed (Participants) | 34 | 65 | 99
scores on a scale
  Week 4, n=34, 65, 99 | -0.3 (0.59) | -0.4 (0.66) | -0.4 (0.63)
  Week 8, n=34, 65, 99 | -0.2 (0.70) | -0.4 (0.71) | -0.4 (0.71)
  Week 12, n=34, 64, 98 | -0.3 (0.62) | -0.4 (0.68) | -0.3 (0.66)
  Week 16, n=34, 62, 96 | -0.3 (0.57) | -0.4 (0.69) | -0.3 (0.65)
  Week 20, n=20, 56, 76 | -0.2 (0.37) | -0.3 (0.67) | -0.3 (0.61)
  Week 24, n=10, 49, 59 | 0.0 (0.00) | -0.3 (0.75) | -0.3 (0.69)

42. Secondary Outcome: Mean Change From Baseline in the Item 6 (Difficult to Do Any Sport) Score of the DLQI at Weeks 4, 8, 12, 16, 20, and 24 in the Second Treatment Phase
Description: as for outcome 19
Time Frame: as for outcome 29
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP | Total
Number analyzed (Participants) | 34 | 65 | 99
scores on a scale
  Week 4, n=34, 65, 99 | -0.3 (0.45) | -0.3 (0.54) | -0.3 (0.51)
  Week 8, n=34, 65, 99 | -0.2 (0.52) | -0.3 (0.56) | -0.3 (0.55)
  Week 12, n=34, 64, 98 | -0.2 (0.46) | -0.3 (0.60) | -0.2 (0.55)
  Week 16, n=34, 62, 96 | -0.2 (0.48) | -0.3 (0.57) | -0.2 (0.54)
  Week 20, n=20, 56, 76 | -0.2 (0.37) | -0.3 (0.53) | -0.3 (0.49)
  Week 24, n=10, 49, 59 | -0.2 (0.63) | -0.2 (0.54) | -0.2 (0.55)

43. Secondary Outcome: Mean Change From Baseline in the Item 7 (Problem at Work or Studying) Score of the DLQI at Weeks 4, 8, 12, 16, 20, and 24 in the Second Treatment Phase
Description: as for outcome 20
Time Frame: as for outcome 29
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP | Total
Number analyzed (Participants) | 34 | 65 | 99
scores on a scale
  Week 4, n=34, 65, 99 | -0.3 (0.51) | -0.6 (0.83) | -0.5 (0.75)
  Week 8, n=34, 65, 99 | -0.2 (0.65) | -0.5 (0.85) | -0.4 (0.80)
  Week 12, n=34, 64, 98 | -0.1 (0.56) | -0.5 (0.93) | -0.4 (0.83)
  Week 16, n=34, 62, 96 | -0.2 (0.43) | -0.5 (0.84) | -0.4 (0.74)
  Week 20, n=20, 56, 76 | -0.2 (0.37) | -0.4 (0.78) | -0.4 (0.71)
  Week 24, n=10, 49, 59 | -0.1 (0.57) | -0.4 (0.91) | -0.4 (0.87)

44. Secondary Outcome: Mean Change From Baseline in the Item 8 (Problem With Partner/Friends) Score of the DLQI at Weeks 4, 8, 12, 16, 20, and 24 in the Second Treatment Phase
Description: as for outcome 21
Time Frame: as for outcome 29
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP | Total
Number analyzed (Participants) | 34 | 65 | 99
scores on a scale
  Week 4, n=34, 65, 99 | 0.0 (0.00) | -0.2 (0.49) | -0.1 (0.40)
  Week 8, n=34, 65, 99 | 0.0 (0.17) | -0.2 (0.51) | -0.1 (0.43)
  Week 12, n=34, 64, 98 | 0.0 (0.17) | -0.2 (0.41) | -0.1 (0.45)
  Week 16, n=34, 62, 96 | 0.0 (0.17) | -0.2 (0.52) | -0.1 (0.44)
  Week 20, n=20, 56, 76 | 0.1 (0.22) | -0.1 (0.41) | -0.1 (0.38)
  Week 24, n=10, 49, 59 | 0.2 (0.63) | -0.1 (0.58) | -0.1 (0.60)

45. Secondary Outcome: Mean Change From Baseline in the Item 9 (Caused Any Sexual Difficulties) Score of the DLQI at Weeks 4, 8, 12, 16, 20, and 24 in the Second Treatment Phase
Description: as for outcome 22
Time Frame: as for outcome 29
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP | Total
Number analyzed (Participants) | 34 | 65 | 99
scores on a scale
  Week 4, n=34, 65, 99 | -0.1 (0.29) | -0.1 (0.43) | -0.1 (0.39)
  Week 8, n=34, 65, 99 | -0.1 (0.24) | -0.2 (0.44) | -0.1 (0.39)
  Week 12, n=34, 64, 98 | -0.1 (0.24) | -0.2 (0.49) | -0.1 (0.42)
  Week 16, n=34, 62, 96 | -0.1 (0.24) | -0.2 (0.50) | -0.1 (0.43)
  Week 20, n=20, 56, 76 | -0.1 (0.22) | -0.2 (0.46) | -0.1 (0.41)
  Week 24, n=10, 49, 59 | 0.0 (0.00) | -0.1 (0.46) | -0.1 (0.42)

46. Secondary Outcome: Mean Change From Baseline in the Item 10 (Problem Caused by Skin Treatment) Score of the DLQI at Weeks 4, 8, 12, 16, 20, and 24 in the Second Treatment Phase
Description: as for outcome 23
Time Frame: as for outcome 29
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP | Total
Number analyzed (Participants) | 34 | 65 | 99
scores on a scale
  Week 4, n=34, 65, 99 | -0.1 (0.50) | -0.3 (0.59) | -0.2 (0.56)
  Week 8, n=34, 65, 99 | -0.1 (0.36) | -0.3 (0.62) | -0.2 (0.55)
  Week 12, n=34, 64, 98 | 0.0 (0.30) | -0.3 (0.60) | -0.2 (0.52)
  Week 16, n=34, 62, 96 | -0.1 (0.29) | -0.2 (0.73) | -0.2 (0.62)
  Week 20, n=20, 56, 76 | -0.1 (0.31) | -0.2 (0.69) | -0.2 (0.61)
  Week 24, n=10, 49, 59 | 0.1 (0.32) | -0.2 (0.73) | -0.1 (0.68)

47. Secondary Outcome: Participant's Global Assessment of Treatment Satisfaction in the Second Treatment Phase
Description: Participant's global assessment of treatment satisfaction is a method used to evaluate a participant's treatment satisfaction. Participants rated any improvement or worsening of their symptoms compared to Baseline by using the following 9-point scale: +4, Complete abolishment of signs and symptoms; +3, Marked improvement; +2, Moderate improvement; +1, Slight improvement; 0, Unchanged; -1, Slight worsening; -2, Moderate worsening; -3, Marked worsening; and -4, Very marked worsening.
Time Frame: Weeks 4 (Study Week 20 to Week 28), 8 (Study Week 24 to 32), 12 (Study Week 28 to 36), 16 (Study Week 32 to 40), 20 (Study Week 36 to 40), and 24 (Study Week 40) in the Second Treatment Phase
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP | Total
Number analyzed (Participants) | 34 | 65 | 99
scores on a scale
  Week 4, n=34, 65, 99 | 3.2 (0.88) | 2.8 (1.10) | 2.9 (1.04)
  Week 8, n=34, 65, 99 | 3.0 (1.14) | 2.8 (1.09) | 2.9 (1.11)
  Week 12, n=34, 64, 98 | 2.8 (1.14) | 2.7 (1.27) | 2.7 (1.22)
  Week 16, n=34, 62, 96 | 2.6 (1.35) | 2.6 (1.36) | 2.6 (1.35)
  Week 20, n=20, 56, 76 | 2.3 (1.29) | 2.3 (1.46) | 2.3 (1.41)
  Week 24, n=10, 49, 59 | 1.7 (1.34) | 2.1 (1.52) | 2.0 (1.49)

48. Secondary Outcome: Duration of Effect
Description: Duration of effect is defined as the number of days between the date of first treatment and the date of the first recording of >50% production in gravimetric assessment compared to Baseline.
Time Frame: Up to Week 40
Population: FAS1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP
Number analyzed (Participants) | 78 | 74
days | 273.0 [171.0 to NA] — The upper limit of the 95% CI for the median cannot be estimated because the follow-up duration is limited. | 35.0 [28.0 to 56.0]

ADVERSE EVENTS:
Description: The number of participants at risk in the BTX arm includes the participants who received at least one BTX treatment in either the First or Second Treatment Periods. The number of participants at risk in the placebo arm includes the participants who received at least one dose of placebo in the First Treatment Period.
Arm/Group | BTX 50 U in First and Second TPs | Placebo in First TP; BTX 50 U in Second TP
Serious Adverse Events (participants affected / at risk) | 1/144 | 1/74
Other Adverse Events (participants affected / at risk) | 23/144 | 9/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BTX 50 U in First and Second TPs (N=144) | Placebo in First TP; BTX 50 U in Second TP (N=74)
Colitis (Gastrointestinal disorders) | 0 | 1
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BTX 50 U in First and Second TPs (N=144) | Placebo in First TP; BTX 50 U in Second TP (N=74)
Nasopharyngitis (Infections and infestations) | 23 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.